CLINICAL TRIAL: NCT03890991
Title: Self-Care for Older People With Diabetes Mellitus (SCOPE-DM): Live Well With Diabetes Programme
Brief Title: Self-Care for Older People With Diabetes Mellitus
Acronym: SCOPE-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Tsao Foundation Singapore (Unknown)
Responsible Party: Principal Investigator, Raymond Boon Tar Lim, Lecturer, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-18-074
Record Dates: First submitted 2019-03-14; First posted 2019-03-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Intervention; Self-efficacy; Diabetes Self-care Activities; Self-Monitoring of Blood Glucose; Diabetes; Community; Older people with diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCOPE-DM only (Experimental): Participation in SCOPE-DM programme without supply of glucometers and accessories
  Interventions: Behavioral: SCOPE-DM
- SCOPE-DM with 3 months' supply of glucometer (Active Comparator): Participation in SCOPE-DM programme with 3 months' supply of glucometers and accessories
  Interventions: Behavioral: SCOPE-DM with 3 months' supply of glucometer
- SCOPE-DM with 6 months' supply of glucometer (Active Comparator): Participation in SCOPE-DM programme with 6 months' supply of glucometers and accessories.
  Interventions: Behavioral: SCOPE-DM with 6 months' supply of glucometer
- Control (No Intervention): Usual care by healthcare provider/ clinics of Tsao Foundation without participation in SCOPE-DM programme

INTERVENTIONS:
Behavioral: SCOPE-DM — The 12-week programme aims to support motivation and enable capability for managing diabetes. To this end, the sessions will integrate the knowledge and practical skills components offered in traditional diabetes education with psychological techniques and principles for behavioural change: problem solving, goal-setting and monitoring. The programme offers the potential for older people to learn about their condition and treatment in a psychologically-motivating and confidence-enhancing structure - as such the emphasis is on empowering individuals to make choices and lifestyle changes in line with treatment recommendations through the use of problem solving, goal setting and feedback, and not just on knowledge transfer which has not been shown to be successful in behavioural change. The content and delivery format will largely be informed by motivational interviewing
  Arms: SCOPE-DM only
Behavioral: SCOPE-DM with 3 months' supply of glucometer — Participants in this arm will participate in the SCOPE-DM programme and use the glucometer for 3 months.
  Arms: SCOPE-DM with 3 months' supply of glucometer
Behavioral: SCOPE-DM with 6 months' supply of glucometer — Participants in this arm will participate the in SCOPE-DM programme and use the glucometer for 6 months.
  Arms: SCOPE-DM with 6 months' supply of glucometer

SUMMARY:
In Singapore, the prevalence of diabetes was approximately 12.8% in 2014 and was projected to rise to 22.7% in 2035. In 2015, the International Diabetes Federation (IDF) reported that Singapore has the second highest proportion of diabetic patients among developed nations. The impact of poorly controlled diabetes on the individual, family and health system is well known. Previous studies have shown that older persons, specifically those with chronic conditions such as diabetes, often lack sufficient knowledge about their condition and thus frequently have poor self-management skills, which is essential for good health outcome.

Health education among older persons, particularly those with chronic illnesses, has long been promoted as a priority. Chodosh and colleagues (2005) determined that there were benefits and significant improvement in blood glucose and blood pressure for chronic disease self-management programs for older adults with diabetes and high blood pressure respectively in a meta-analysis study. This project [Self-Care for Older People with Diabetes Mellitus (SCOPE-DM)] was therefore developed to help community-dwelling older patients with type 2 diabetes to effectively manage their disease by reducing diabetes-related risk factors and complications, leading to an improvement in their psychological well-being and health-related quality of life, as well as a reduction in future healthcare requirements from family and society. This study aims to investigate the effectiveness of the SCOPE-DM programme in improving the self-efficacy, motivation, medication adherence, health-related quality of life and diabetes knowledge among community-dwelling older adults with type 2 diabetes in Singapore.

This proposed study is a prospective, four-group cluster randomized controlled trial. The participants will be followed up for 6 months at the community sites and Hua Mei Clinics of the Tsao Foundation. A set of questionnaires will be used to assess participants' self-efficacy, diabetic self-care activities, health-related quality of life (HRQoL), diabetes knowledge and medication adherence. Process evaluation will also be conducted to assess the acceptability, strengths and weaknesses of the 'SCOPE-DM: Live Well with Diabetes' programme based on the participants' perspectives through the conduct of qualitative interviews.

DETAILED DESCRIPTION:
Overview

This study is a prospective, four-group cluster randomized controlled trial. The participants will be followed up for 6 months at the community sites or Hua Mei Clinics of the Tsao Foundation.

The 4 groups are:

i. Control group receiving routine care from their healthcare provider/ clinics of Tsao Foundation

ii. Intervention group 1 receiving the SCOPE-DM programme without supply of glucometers and accessories

iii. Intervention group 2 receiving the SCOPE-DM programme as well as 3 months' supply of glucometers and accessories

iv. Intervention group 3 receiving the SCOPE-DM programme as well as 6 months' supply of glucometers and accessories

A staff of Tsao Foundation will recruit community-dwelling adults with diabetes from the 68 community sites around Singapore. After which, the research associate (RA) or Fellow appointed to represent the Site Principal Investigator will screen the individuals participating for eligibility to join this research study. Alternatively, potential participants will be referred to the RA or Fellow to be screened for eligibility. Eligible individuals will be invited to participate in the research study, of which interested individuals will be explained with the study procedure and informed consent will be taken by the RA.

Inclusion Criteria:

* Individuals with type 2 diabetes mellitus
* Aged 55 to 99 years old (both inclusive)
* Community-dwelling

Exclusion Criteria:

* Individuals with Type 1 diabetes mellitus
* Unable to communicate independently in English or Mandarin
* Mentally incapacitated individuals

The 68 sites will form the cluster sites for the study and will be assigned to any one of the 4 groups via a randomisation process (control, intervention group 1, 2 and 3). The randomisation process will be generated by the research team before recruitment begins using a computerised programme. Each group will thus consist of 17 sites. All the participants belonging to each group of 17 sites will be invited to participate in the study if they meet the inclusion criteria until we have reached the target number of 80 for each group.

Questionnaire administration

Questionnaires to elucidate the humanistic outcomes will be administered at baseline, 3 and 6 months from baseline respectively for all 4 groups. Each questionnaire administration will last for around 45 minutes.

The questionnaire will be used to assess participants' self-efficacy, diabetic self-care activities, health-related quality of life (HRQoL), diabetes knowledge and medication adherence. Participant demographics, anthropometric parameters, past medical history, and current medication use will be collected. A staff from Tsao Foundation will provide the clinical data and laboratory test results (HbA1c, blood pressure, TChol, LDL-C, HDL-C, TG, BMI and adherence to yearly eye and foot screenings) to the RA or Fellow of the project. Consent will be obtained from the participants before Tsao Foundation releases the clinical data and laboratory test results to the research team. The data and test results will be printed out by the staff of Tsao Foundation and handed over to the RA or Fellow in an opaque sealed envelope. Only the RA or Fellow, Co-Investigators and Principal Investigators of the study are authorised to open the sealed envelope and retrieve data. A representative of Tsao Foundation may call the subject for care- and administrative-related matters if needed such as reminding the participants to attend the SCOPE-DM programme or to follow up on the questionnaire administration.

Process Evaluation

The purpose of the process evaluation is to assess the acceptability, strengths and weaknesses of the 'SCOPE-DM: Live Well with Diabetes' programme based on the participants' perspectives. A qualitative approach using individual face-to-face audio-recorded interviews will be adopted. The RA will conduct these interviews after the completion of the study intervention and upon the participant's consent. A purposive sample of 30 participants will be recruited from intervention groups to participate in the interviews to share their experiences while in the programme as well as obtain their opinions and suggestions to improve the programme.

All interviews will be audio-recorded. An interview guide will be developed based on the overall aim of the SCOPE-DM program. The participants will be reminded not to reveal any information that may identify themselves before the interview commences as interviews will be audio-recorded. The qualitative interview will last for about 1 hour.

The administration of the questionnaires and conduct of the interviews will be done at a room with privacy and confidentiality maintained at the Hua Mei Clinics or any of the community sites. The venue to administer the questionnaires and interviews are appropriately equipped with tables, chairs and rooms to ensure the privacy and confidentiality of participants.

Details of SCOPE-DM intervention programme

Tsao Foundation's trained diabetes nurse educators will commence the SCOPE-DM intervention programme once 8 to 10 participants agreed to participate. Tsao Foundation will be responsible for training 20 diabetes nurse educators to deliver the programme. The SCOPE-DM programme will be conducted at Hua Mei Clinics or any of the community sites. Each session will last around 2 hours.

The programme aims to support motivation and enable capability for managing diabetes. To this end, the session will integrate the knowledge and practical skills components offered in traditional diabetes education with psychological techniques and principles for behavioural change: problem solving, goal-setting and monitoring. The programme offers the potential for older people to learn about their condition and treatment in a psychologically-motivating and confidence-enhancing structure - as such the emphasis is on empowering individuals to make choices and lifestyle changes in line with treatment recommendations through the use of problem solving, goal setting and feedback, and not just on knowledge transfer which has not been shown to be successful in behavioural change. The content and delivery format will largely be informed by motivational interviewing (MI).

Motivational interviewing is a well-recognized person-centered counselling approach aiming at eliciting and strengthening motivation to change. It is designed to guide towards a specific goal by eliciting and exploring the person's own reasons for change, goals and values within an atmosphere of acceptance and empathy.There is now a wealth of evidence from randomized trials for the effectiveness of MI in health behavioural change.To facilitate engagement and rapport with the participants, MI will be blended with guided autobiography as means to share life experiences and meaning and hence allowing for better alignment of health behavioural changes with participants' personal goals and values.

The 2-hour weekly sessions will apply the strategies of group-based activities, problem solving, motivational building and goal setting, vicarious experience, enactive attainment and physiological feedback. Themes will include dealing with the medical management of the disease (medical management); maintaining, changing, and creating new meaningful behaviours or life roles (role management), and dealing with the emotional consequences of having a chronic condition (emotional management).

These topics are taught by means of skills mastery through goal setting and feedback on progress, modelling of self-management behaviours and problem-solving strategies, and social persuasion through group support and guidance for individual self-management efforts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes mellitus
* Aged 55 to 99 years old (both inclusive)
* Community-dwelling

Exclusion Criteria:

* Individuals with Type 1 diabetes mellitus
* Unable to communicate independently in English or Mandarin
* Mentally incapacitated individuals

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy assessed using the General Self-efficacy Scale | 6 months
  Participants' level of self-efficacy is assessed using the ten-item General Self-efficacy Scale. Participants indicate their responses on a Likert scale of 1 ("Not at all true") to 4 ("Exactly true"). Scores for the ten items are then summed, with higher summed scores indicating higher levels of self-efficacy. The minimum possible summed score is 10 and the maximum possible summed score is 40. Participants in the three intervention conditions are hypothesized to have statistically significantly higher summed scores post-intervention, compared to control condition participants.
Diabetes self-care activities measured using the Revised Summary of Diabetes Self-care Activities | 6 months
  Diabetes self-care activities are assessed using a 13-item scale. Participants indicate their responses to items 1 to 12 on a scale of 0 to 7 corresponding to the number of days within the past seven days that they have performed the activities indicated. For item 13, participants indicate whether they have smoked within the past seven days, and if so, how many cigarettes on an average day. For each regimen area of general diet, exercise, blood sugar testing, footcare, and medications, the responses of the corresponding items are averaged to indicate the mean number of days, with a higher value indicating a higher level of self-care activity for the regimen area. A score of 0 is assigned to non-smoking and a score of 1 assigned to smoking, with higher scores indicating lower self-care. Participants in the three intervention conditions are hypothesized to have a statistically significantly higher level of self-care activities post-intervention, compared to control participants.

SECONDARY OUTCOMES:
Diabetes-specific quality of life measured using the Audit of Diabetes-Dependent Quality of Life | 6 months
  The first two items ask participants about current quality of life (rated on a 7-point Likert Scale ranging from -3 to +3) and diabetes-dependent quality of life (rated on a 5-point Likert scale ranging from -3 to +1. Lower scores indicate a lower quality of life. The subsequent 19 items assess the impact of diabetes on 19 life domains. For each life domain, participants indicate the level of impact on a 5-point Likert scale ranging from -3 ("greatest") to +1 ("least"), and the importance of the domain to them on a 4-point Likert scale ranging from 3 ("very important") to 0 ("Not at all important"). The two ratings for each item are then multiplied before the products are averaged across all applicable domains for an average weighted impact score ranging from -9 to 3. Scores equal to or above the lower quartile score indicate a higher quality of life. The outcome measure will be the proportion of participants in each condition with scores equal or above the lower quartile score.
Participants' level of knowledge of Diabetes assessed using the Revised Michigan Diabetes Knowledge Questionnaire | 6 months
  Participants' level of knowledge of Diabetes is assessed using the 20-item Revised Michigan Diabetes Knowledge Questionnaire (Diabetes Knowledge Test). Participants indicate their responses from the options of "True", "False" or "Don't know". A higher proportion of correct responses on this scale is indicative of a higher level of knowledge regarding Diabetes. Participants in the three intervention conditions are hypothesized to have statistically significantly higher levels of knowledge regarding Diabetes post-intervention, compared to control condition participants.
Participants' level of medication adherence assessed using Medication Adherence Report Scale | 6 months
  Level of medication adherence is assessed using the five-item Medication Adherence Report Scale. Participants indicate their responses on a five-point Likert scale ranging from 1 ("Always") to 5 ("Never"). Higher scores are indicative of higher levels of medication adherence, with a minimum possible summed score of 5 and a maximum possible summed score of 25. The target score is 25 indicating perfect adherence to medication, and the outcome measure would be the proportion of participants in each study condition with a summed score of 25.
Proportion of participants with optimal Glycated haemoglobin Level (HbA1c Level) of 7% or lower | 6 months
  Glycated haemoglobin level is an indication of an individual's average blood glucose level over the past three months. For individuals with type 2 diabetes, in general, the optimal HbA1c level should be 7% or lower. Thus, the outcome measured would be the proportion of participants from each study condition with Glycated haemoglobin level of 7% or lower.
Proportion of participants with optimal Systolic and Diastolic Blood Pressure | 6 months
  The optimal Systolic and Diastolic Blood Pressure would be below 140 over 80mmHg. Thus, the outcome measured would be the proportion of participants from each study condition with Systolic and Diastolic Blood Pressure below 140 over 80mmHg.
Proportion of participants with optimal levels of Total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglyceride | 6 months
  The outcome measured would be the proportion of participants from each study condition with the optimal levels of Total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglyceride. Optimal level for total cholesterol should be less than 5.2mmol/L, optimal high-density lipoprotein cholesterol level should be more than 1.5mmol/L, optimal low-density lipoprotein cholesterol level should be less than 2.6 mmol/L and optimal triglyceride level should be less than 1.7mmol/L.
Proportion of participants with optimal Body Mass Index between 18.5 and 22.9 | 6 months
  The outcome measured would be the proportion of participants from each study condition with optimal Body Mass Index between 18.5 and 22.9 (both inclusive).
Proportion of participants who adhere to yearly eye and foot screening | 6 months
  The outcome measured would be the proportion of participants from each study condition with self-reported adherence to yearly eye screening and foot screening. Yearly eye screening and foot screening are assessed through two of the items in the questionnaire asking participants if they have gone for yearly eye screening and foot screening respectively. For both items, response options are "Yes" or "No". Participants who answer "Yes" to both questions would be regarded as having adhered to yearly eye and foot screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Whampoa Community Club, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No